CLINICAL TRIAL: NCT05345483
Title: REscue Stenting With CREDO® Heal for Recanalisation After Unsuccessful Thrombectomy (RECHRUT)
Acronym: RECHRUT
Status: Recruiting | Type: Observational
Sponsor: Acandis GmbH (Industry)
Responsible Party: Sponsor
Other Study IDs: RECHRUT
Record Dates: First submitted 2022-04-07; First posted 2022-04-26 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Rescue Stenting

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Rescue stenting with CREDO heal Stent together with NeuroSpeed PTA Balloon Catheter — Rescue stenting with CREDO heal Stent together with NeuroSpeed PTA Balloon Catheter

SUMMARY:
Goal of the study is to evaluate the efficacy and safety of acute permanent stenting of symptomatic intracranial stenosis following unsuccessful recanalization by thrombectomy in acute ischemic stroke with large vessel occlusion using the self-expandable CREDO® heal Stent.

ELIGIBILITY:
Inclusion Criteria:

* Patients, treated with CREDO® heal according to IFU
* Over 18 years old
* With acute persistent vascular occlusion due to high grade intracranial artery stenosis in the anterior or posterior circulation for which alternative therapy concepts are not considered or fail
* With suspected underlying stenosis of the occluded artery, which is suitable for PTA and stenting according to the treating physician's assessment and/or persistent occlusion after failed recanalization by mechanical thrombectomy of the target region
* With small to moderate infarct core prior to initiation of thrombectomy (CT ASPECTS 6-10, DWI lesion < 70 ml)
* With symptoms onset less than 24 hours before start of the procedure
* Treated with study device following at least one futile mechanical recanalization attempt with a stent retriever, direct aspiration or combination of both
* With pre-stroke disability mRS 0-2

Exclusion Criteria:

* Any contraindication according to IFU and patients:
* With atherosclerotic (probable according to clinical, anamnestic or laboratory chemical testing) vessel constrictions (high-grade intracranial stenoses > 70 %) with significant circulatory disturbance (haemodynamic infarct pattern and signs of restricted collaterals) and recurrent symptoms in spite of medical therapy
* With contraindication against treatment with anti-platelet medication
* Participating in another trial

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients who were treated with CREDO® heal due to acute ischemic stroke and proven occlusion with unsuccessful recanalization after endovascular treatment with mechanical thrombectomy and suspected underlying stenosis of the occluded intracranial artery, which is suitable to PTA and stenting based on the decision of the treating physician.
Sampling Method: Non-Probability Sample
Enrollment: 153 (Estimated)
Dates: Start 2023-01-25 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Primary Technical Efficacy Endpoint- proportion of patients with eTICI 2b-3 at the end of the treatment procedure. | Assessed at the end of the treatment procedure.
  • Technical success defined as successful recanalization of the occluded vessel (expanded treatment in cerebral ischemia score (eTICI) of 2b-3) at the end of the procedure.
Primary Clinical Efficacy Endpoint- proportion of patients with mRS 0-2 at 90 (± 20) days after procedure. | 90 (± 20) days.
  • Good clinical outcome 90 (± 20) days after stroke defined as a score of 0-2 on the modified Ranking Scale (mRS 0-2).

CONTACTS AND LOCATIONS:
Locations (17):
- Germany (17):
  - Institut für Radiologie und Neuroradiologie, Klinikum Aschaffenburg-Alzenau, Aschaffenburg
  - Klinik für Diagnostische Radiologie und Neuroradiologie; Universitätsklinikum Augsburg, Augsburg
  - Klinik für Diagnostische und Interventionelle Neuroradiologie; Universitätsklinikum Bonn, Bonn
  - Institut für Diagnostische und Interventionelle Radiologie, Neuroradiologie und Nuklearmedizin, Klinikum Bremerhaven-Reinkenheide, Bremerhaven
  - Institut und Poliklinik für Diagnostische und Interventionelle Neuroradiologie, Universitätsklinikum Dresden, Dresden
  - Klinik für Radiologie und Neuroradiologie, Sana Klinikum, Duisburg
  - Diagnostische und interventionelle Radiologie, Helios Klinikum Erfurt, Erfurt
  - Diagnostische und Interventionelle Neuroradiologie, Universitätsmedizin Halle, Halle
  - Abteilung für Radiologie, Neuroradiologie und Nuklearmedizin, Asklepios Klinikum Altona, Hamburg
  - Klinik und Poliklinik für Neuroradiologische Diagnostik und Intervention, Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Radiologie / Neuroradiologie, Askleopis Klinik St. Georg, Hamburg
  - Klinik für Neuroradiologie, Westpfalz-Klinikum, Kaiserslautern
  - Abteilung für Radiologie und Nuklearmedizin, Sana Kliniken, Lübeck
  - Interventionelle Neuroradiologie, Universitätsklinikum Münster, Münster
  - Institut für Radiologie und Neuroradiologie, Evangelisches Krankenhaus Oldenburg, Oldenburg
  - Klinik für Radiologie, Neuroradiologie und Nuklearmedizin, Klinikum Vest, Recklinghausen
  - Institut für Diagnostische und Interventionelle Neuroradiologie, Städtisches Klinikum, Solingen

IPD SHARING:
Plan to Share IPD: No